CLINICAL TRIAL: NCT00654901
Title: Immunogenicity Study of the Antibody Persistence and Booster Effect of the DTaP-IPV-Hep B-PRP~T Combined Vaccine at 15 to 18 Months of Age Following a Primary Series of DTaP-IPV-Hep B-PRP~T or Infanrix Hexa™ Administered at 2, 4, and 6 Months of Age in Healthy Mexican Infants
Brief Title: Study of the DTaP-IPV-Hep B-PRP~T Combined Vaccine Following a Primary Series of DTacP IPV-HepB-PRP-T or Infanrix Hexa™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L21
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis; Haemophilus Influenzae Type B Infection
Keywords: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis; Invasive Haemophilus influenzae type b.; Haemophilus Influenzae Type B Infection
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DTaP-IPV-Hep B-PRP~T Batch 1 (Experimental): Participants had received 3 primary doses of Batch 1 of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) in Study A3L11 (NCT00404651); and will receive a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
  Interventions: Biological: DTaP-IPV-Hep B-PRP~T vaccine (Batch 1)
- DTaP-IPV-Hep B-PRP~T Batch 2 (Experimental): Participants had received 3 primary doses of Batch 1 of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) in Study A3L11 (NCT00404651) and will receive a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
  Interventions: Biological: DTaP-IPV-Hep B-PRP~T vaccine (Batch 2)
- DTaP-IPV-Hep B-PRP~T Batch 3 (Experimental): Participants had received 3 primary doses of Batch 1 of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) in Study A3L11 (NCT00404651) and will receive a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
  Interventions: Biological: DTaP-IPV-Hep B-PRP~T vaccine (Batch 3)
- Infanrix Hexa™ (Active Comparator): Participants had received 3 primary doses of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), (Infanrix Hexa™) plus Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed in Study A3L11 (NCT00404651) and received a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
  Interventions: Biological: Infanrix Hexa™

INTERVENTIONS:
Biological: DTaP-IPV-Hep B-PRP~T vaccine (Batch 1) — 0.5 mL, Intramuscular
  Arms: DTaP-IPV-Hep B-PRP~T Batch 1
Biological: DTaP-IPV-Hep B-PRP~T vaccine (Batch 2) — 0.5 mL, Intramuscular
  Arms: DTaP-IPV-Hep B-PRP~T Batch 2
Biological: DTaP-IPV-Hep B-PRP~T vaccine (Batch 3) — 0.5 mL, Intramuscular
  Arms: DTaP-IPV-Hep B-PRP~T Batch 3
Biological: Infanrix Hexa™ — 0.5 mL, Intramuscular
  Arms: Infanrix Hexa™

SUMMARY:
This is a follow-up of Study A3L11 (NCT00404651).

Immunogenicity

* To describe the antibody persistence following a primary series vaccination of either DTaP-IPV-Hep B-PRP~T or Infanrix hexa™.
* To describe the immunogenicity of a booster dose of DTaP-IPV-HepB-PRP~T in a subset of subjects.

Safety

- To describe the safety profile after a booster dose of DTacP-IPV-HepB-PRP~T.

ELIGIBILITY:
Inclusion Criteria:

* Toddlers previously included in Study A3L11 (NCT00404651) who completed the three-dose primary series vaccination of either DTaP-IPV-HepB-PRP-T or Infanrix hexa™ at 2, 4 and 6 months of age
* Toddlers of 15 to 18 months (456 to 578 days) of age, inclusive
* Informed Consent Form signed by at least one parent or legal representative and two mandatory witnesses
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the booster vaccination.
* Planned participation in another clinical trial during the present trial period.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroid therapy.
* Systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to a vaccine containing the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the last 3 months.
* Any vaccination in the 4 weeks preceding the booster vaccination.
* Any vaccination planned until the next visit.
* History of documented pertussis, tetanus, diphtheria, polio, Haemophilus influenzae type b or hepatitis B (HB) infection(s) (confirmed either clinically, serologically or microbiologically).
* Administration of a vaccine against pertussis, tetanus, diphtheria, polio, Hib, and/or hepatitis B infection(s) since the end of participation in Study A3L11.
* Coagulopathy, thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination.
* Known maternal history of human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbsAg) or Hepatitis C seropositivity.
* Subjects with any related serious adverse event that occurred following the three-dose primary series administration of the investigational vaccine or of the reference vaccine in Study A3L11.
* History of seizures.
* Febrile (temperature ≥38.0°C) or acute illness on the day of inclusion
* Known contraindication to further vaccination with a pertussis vaccine, i.e.: Encephalopathy; Temperature >40.0°C within 48 hours following a vaccine injection, not due to another identifiable cause during the primary series; Inconsolable crying that occurred for >3 hours within 48 hours following vaccine injection during the primary series; Hypotonic hyporesponsive episode within 48 hours following vaccine injection during the primary series; Seizures with or without fever within 3 days following vaccine injection.

Ages: 15 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 881 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (4):
- Mexico (4):
  - Estado de México
  - Insurgentes Cuicuilco
  - Monterrey
  - Puebla City

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 25 March 2008 to 28 November 2008 at 5 clinical centers in Mexico.
Pre-assignment Details: A total of 881 participants who met the inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- DTaP-IPV-Hep B-PRP~T Batch 1: Participants had received 3 primary doses of Batch 1 of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) in Study A3L11 and received a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
- DTaP-IPV-Hep B-PRP~T Batch 2: Participants had received 3 primary doses of Batch 2 of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) in Study A3L11 and received a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
- DTaP-IPV-Hep B-PRP~T Batch 3: Participants had received 3 primary doses of Batch 3 of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) in Study A3L11 and received a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
- Infanrix Hexa™: Participants had received 3 primary doses of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), (Infanrix hexa™), plus Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed in Study A3L11 and received a booster dose of DTaP-IPV-Hep B-PRP~T at Day 0 in the present study.
Period: Overall Study
Arm/Group | DTaP-IPV-Hep B-PRP~T Batch 1 | DTaP-IPV-Hep B-PRP~T Batch 2 | DTaP-IPV-Hep B-PRP~T Batch 3 | Infanrix Hexa™
Started | 254 | 262 | 252 | 113
Completed | 250 | 262 | 250 | 113
Not Completed | 4 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- DTaP-IPV-Hep B-PRP~T Batch 1: Participants had received 3 primary doses of Batch A of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) in Study A3L11 and received a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
- DTaP-IPV-Hep B-PRP~T Batch 2: Participants had received 3 primary doses of Batch B of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-Hep B-PRP~T) in Study A3L11 and received a booster dose of (DTaP-IPV-Hep B-PRP~T) at Day 0 in the present study.
- Infanrix Hexa™: Participants had received 3 primary doses of Diphtheria (D), Tetanus (T), Pertussis (acellular, component [aP]), Hepatitis B (Hep B, [recombinant DNA]) and poliomyelitis (Inactivated [IPV]) (Infanrix hexa™), plus Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed in Study A3L11 and received a booster dose of DTaP-IPV-Hep B-PRP~T at Day 0 in the present study.
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV-Hep B-PRP~T Batch 1 | DTaP-IPV-Hep B-PRP~T Batch 2 | DTaP-IPV-Hep B-PRP~T Batch 3 | Infanrix Hexa™ | Total
Number analyzed (Participants) | 254 | 262 | 252 | 113 | 881
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 254 | 262 | 252 | 113 | 881
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17.3 (1.51) | 17.2 (1.47) | 17.4 (1.42) | 17.1 (1.51) | 17.3 (1.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 125 | 130 | 58 | 438
  Male | 129 | 137 | 122 | 55 | 443
Region of Enrollment [Number; unit: Participants]
  Mexico | 254 | 262 | 252 | 113 | 881

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of Antibodies Before and After Booster Vaccination With DTaP-IPV-Hep B-PRP~T
Description: Antibody titers were measured for hepatitis B (Hep B) by enhanced chemiluminescence detection, for Haemophilus influenzae type b (PRP) by Farr type radioimmunoassay, for diphtheria by toxin neutralization test, and for tetanus by enzyme linked immunosorbent assay (ELISA). Antibody titers were measured for poliovirus types 1, 2, and 3 by neutralization assay. Antibody titers were measured for pertussis toxoid (PT) and filamentous hemagglutinin (FHA) by ELISA.
Time Frame: Day 0 (pre-booster) and Day 30 (one month post-booster)
Population: Geometric mean titers were assessed in a subset of participants with endpoint data who did not have any protocol deviation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV-Hep B-PRP~T Batch 1 | DTaP-IPV-Hep B-PRP~T Batch 2 | DTaP-IPV-Hep B-PRP~T Batch 3 | Infanrix Hexa™
Number analyzed (Participants) | 58 | 61 | 58 | 65
Titers
  Anti Hep B Pre-booster (N = 58, 60, 58, 65) | 91.1 [56.8 to 146] | 127 [83.9 to 193] | 69.2 [42.3 to 113] | 127 [86.2 to 186]
  Anti Hep B Post-booster (N = 58, 61, 58, 65) | 2167 [1314 to 3573] | 3998 [2510 to 6368] | 1877 [1152 to 3058] | 4757 [3124 to 7243]
  Anti PRP Pre-booster (N = 58, 60, 57, 65) | 1.09 [0.644 to 1.86] | 1.32 [0.937 to 1.87] | 0.880 [0.510 to 1.52] | 1.33 [0.839 to 2.10]
  Anti PRP Post-booster (N = 58, 61, 58, 65) | 64.0 [47.4 to 86.6] | 94.8 [71.6 to 125] | 49.7 [30.6 to 80.6] | 102 [72.8 to 144]
  Anti Diphtheria Pre-booster (N = 58, 60, 57, 64) | 0.116 [0.072 to 0.187] | 0.190 [0.126 to 0.287] | 0.101 [0.062 to 0.164] | 0.081 [0.055 to 0.119]
  Anti Diphtheria Post-booster (N = 58, 61, 58, 65) | 7.78 [4.88 to 12.4] | 15.2 [10.1 to 23.1] | 9.31 [5.80 to 14.9] | 6.01 [3.99 to 9.06]
  Anti Tetanus Pre-booster (N = 58, 60, 57, 65) | 0.330 [0.236 to 0.462] | 0.331 [0.256 to 0.427] | 0.231 [0.167 to 0.318] | 0.297 [0.229 to 0.385]
  Anti Tetanus Post-booster (N = 58, 61, 58, 65) | 5.26 [3.97 to 6.96] | 8.49 [6.50 to 11.1] | 5.55 [4.20 to 7.33] | 6.98 [5.26 to 9.26]
  Anti Polio 1 Pre-booster (N = 57, 59, 57, 65) | 614 [382 to 988] | 663 [458 to 959] | 551 [356 to 853] | 887 [571 to 1378]
  Anti Polio 1 Post-booster (N = 57, 61, 58, 64) | 7037 [4977 to 9949] | 9938 [7418 to 13313] | 8907 [6474 to 12254] | 10173 [7909 to 13086]
  Anti Polio 2 Pre-booster (N = 58, 59, 56, 65) | 936 [584 to 1501] | 839 [530 to 1326] | 531 [309 to 913] | 1267 [747 to 2152]
  Anti Polio 2 Post-booster (N = 56, 61, 58, 64) | 10756 [7636 to 15151] | 10224 [7476 to 13981] | 9232 [6549 to 13014] | 13482 [10245 to 17742]
  Anti Polio 3 Pre-booster (N = 58, 59, 56, 65) | 428 [255 to 719] | 373 [224 to 619] | 241 [130 to 446] | 896 [508 to 1580]
  Anti Polio 3 Post-booster (N = 56, 60, 58, 64) | 6597 [4281 to 10164] | 9575 [6859 to 13365] | 5296 [3503 to 8007] | 13337 [9619 to 18491]
  Anti PT Pre-booster (N = 57, 59, 55, 64) | 15.6 [11.6 to 20.9] | 14.7 [11.8 to 18.4] | 14.5 [11.3 to 18.6] | 15.3 [11.6 to 20.2]
  Anti PT Post-booster (N = 58, 61, 58, 64) | 186 [151 to 230] | 200 [166 to 241] | 171 [137 to 212] | 162 [131 to 200]
  Anti FHA Pre-booster (N = 58, 60, 56, 64) | 42.1 [30.6 to 57.9] | 33.7 [26.0 to 43.8] | 28.3 [21.5 to 37.3] | 25.9 [19.6 to 34.2]
  Anti FHA Post-booster (N = 58, 60, 58, 65) | 410 [336 to 499] | 455 [387 to 536] | 346 [284 to 421] | 291 [242 to 349]

2. Primary Outcome: Number of Participants With Antibody Persistence Before and Immunogenicity Response After Booster Vaccination With DTaP-IPV-Hep B-PRP~T Vaccine
Description: Antibody persistence and immunogenicity response:
  Level 1: ≥ 10 mIU/mL for hepatitis B (Hep B), ≥ 0.15 µg/mL for Haemophilus influenzae type b (PRP), and ≥ 0.01 IU/mL for diphtheria (D) and tetanus (T). Level 2: ≥ 100 mIU/mL (Hep B), ≥ 1.0 µg/mL (PRP), and ≥ 0.1 IU/mL (D and T) Level 3, ≥ 1.0 IU/mL (D and T). Anti-polio titers were defined as ≥ 8 (1.dil), and pertussis toxoid (PT) and filamentous hemagglutinin (FHA) by a 4 fold increase from Day 0.
Time Frame: Day 0 (pre-booster) and Day 30 (one month post-booster)
Population: Antibody persistence and immunogenicity response were assessed in all participants with endpoint data who did not have any protocol deviation that might have interfered with primary criteria evaluation (Per Protocol Population).
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T Batch 1 | DTaP-IPV-Hep B-PRP~T Batch 2 | DTaP-IPV-Hep B-PRP~T Batch 3 | Infanrix Hexa™
Number analyzed (Participants) | 58 | 61 | 58 | 65
Participants
  Anti-Hep B Level 1 Pre-booster (N=58, 60, 58, 65) | 51 | 56 | 51 | 62
  Anti-Hep B Level 2 Pre-booster (N=58, 60, 58, 65) | 29 | 39 | 25 | 38
  Anti-Hep B Level 1 Post-booster (N=58, 61, 58, 65) | 58 | 61 | 57 | 65
  Anti-Hep B Level 2 Post-booster (N=58, 61, 58, 65) | 52 | 58 | 55 | 63
  Anti-PRP Level 1 Pre-booster (N=58, 60, 57, 65) | 51 | 54 | 47 | 60
  Anti-PRP Level 2 Pre-booster (N=58, 60, 57, 65) | 27 | 36 | 25 | 32
  Anti-PRP Level 1 Post-booster (N=58, 61, 58, 65) | 58 | 61 | 58 | 65
  Anti-PRP Level 2 Post booster (N=58, 61, 58, 65) | 58 | 61 | 55 | 64
  Anti-D Level 1 Pre-booster (N=58, 60, 57, 64) | 51 | 59 | 51 | 62
  Anti-D Level 2 Pre-booster (N=58, 60, 57, 64) | 31 | 39 | 29 | 32
  Anti-D Level 1 Post-booster (N=58, 61, 58, 65) | 58 | 60 | 58 | 64
  Anti-D Level 2 Post-booster (N=58, 61, 58, 65) | 56 | 60 | 56 | 63
  Anti-D Level 3 Post-booster (N=58, 61, 58, 65) | 53 | 59 | 53 | 60
  Anti-T Level 1 Pre-booster (N=58, 60, 57, 65) | 58 | 60 | 57 | 65
  Anti-T Level 2 Pre-booster (N=58, 60, 57, 65) | 48 | 52 | 41 | 54
  Anti-T Level 1 Post-booster (N=58, 61, 58, 65) | 58 | 61 | 58 | 65
  Anti-T Level 2 Post-booster (N=58, 61, 58, 65) | 58 | 61 | 58 | 64
  Anti-T Level 3 Post-booster (N=58, 61, 58, 65) | 52 | 58 | 55 | 62
  Anti-Polio 1 Pre-booster (N=57, 59, 57, 65) | 57 | 59 | 57 | 65
  Anti-Polio 1 Post-booster (N=57, 61, 58, 64) | 57 | 61 | 58 | 64
  Anti-Polio 2 Pre-booster (N=58, 59, 56, 65) | 58 | 59 | 56 | 65
  Anti-Polio 2 Post-booster (N=56, 61, 58, 64) | 56 | 61 | 58 | 64
  Anti-Polio 3 Pre-booster (N=58, 59, 56, 65) | 57 | 57 | 53 | 64
  Anti-Polio 3 Post-booster (N=56, 60, 58, 64) | 56 | 60 | 58 | 64
  Anti-PT Post-booster (N=57, 59, 55, 63) | 48 | 57 | 52 | 51
  Anti-FHA Post-booster (N=58, 59, 56, 64) | 48 | 50 | 52 | 57

3. Primary Outcome: Number of Participants With Solicited Injection Site or Systemic Reactions After Vaccination With DTaP-IPV-Hep B-PRP~T Vaccine
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling, Extensive Swelling of Vaccinated Limb. Solicited Systemic Reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia, Irritability.
  Grade 3 reactions were defined as: Pain, cries when injected limb is moved or movement of injected limb reduced; Erythema and swelling, ≥ 5cm; Extensive swelling of limb; Pyrexia, ≥ 39.6ºC; Vomiting ≥ 6 episodes/24 hours or requiring parenteral hydration; Somnolence, sleeping most of time or difficult to wake up; Anorexia, refuses ≥ feeds or most feeds; Irritability, inconsolable.
Time Frame: Days 0 up to 7 after any injection
Population: Solicited reactions were assessed in all subjects who received at least one dose of vaccine, according to the vaccine actually received (Safety Analysis Population).
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T Batch 1 | DTaP-IPV-Hep B-PRP~T Batch 2 | DTaP-IPV-Hep B-PRP~T Batch 3 | Infanrix Hexa™
Number analyzed (Participants) | 254 | 262 | 252 | 113
Participants
  Injection site Pain | 174 | 193 | 177 | 80
  Grade 3 injection site Pain | 8 | 11 | 14 | 6
  Injection site Erythema | 135 | 127 | 135 | 63
  Grade 3 injection site Erythema | 3 | 4 | 5 | 1
  Injection site Swelling | 51 | 69 | 58 | 35
  Grade 3 injection site Swelling | 2 | 3 | 3 | 1
  Extensive Swelling of Vaccinated Limb | 0 | 1 | 0 | 0
  Grade 3 Extensive Swelling of Vaccinated Limb | 0 | 1 | 0 | 0
  Pyrexia | 25 | 35 | 28 | 22
  Grade 3 Pyrexia | 2 | 0 | 2 | 1
  Vomiting | 44 | 49 | 36 | 19
  Grade 3 Vomiting | 0 | 1 | 0 | 1
  Crying | 91 | 91 | 87 | 42
  Grade 3 Crying | 1 | 2 | 2 | 2
  Somnolence | 55 | 66 | 54 | 33
  Grade 3 Somnolence | 5 | 2 | 0 | 0
  Anorexia | 95 | 101 | 87 | 42
  Grade 3 Anorexia | 6 | 5 | 3 | 3
  Irritability | 145 | 166 | 166 | 75
  Grade 3 Irritability | 8 | 3 | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 after the booster injection to up to 6 months post-booster injection.
Arm/Group | DTaP-IPV-Hep B-PRP~T Batch 1 | DTaP-IPV-Hep B-PRP~T Batch 2 | DTaP-IPV-Hep B-PRP~T Batch 3 | Infanrix Hexa™
Serious Adverse Events (participants affected / at risk) | 1/254 | 1/262 | 1/252 | 0/113
Other Adverse Events (participants affected / at risk) | 188/254 | 207/262 | 197/252 | 92/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T Batch 1 (N=254) | DTaP-IPV-Hep B-PRP~T Batch 2 (N=262) | DTaP-IPV-Hep B-PRP~T Batch 3 (N=252) | Infanrix Hexa™ (N=113)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T Batch 1 (N=254) | DTaP-IPV-Hep B-PRP~T Batch 2 (N=262) | DTaP-IPV-Hep B-PRP~T Batch 3 (N=252) | Infanrix Hexa™ (N=113)
Vomiting (Gastrointestinal disorders) | 44 (44) | 49 (49) | 36 (36) | 19 (19)
Solicited Injection Site Erythema (General disorders) | 135 (135) | 127 (127) | 135 (135) | 63 (63)
Solicited Injection Site Pain (General disorders) | 174 (174) | 193 (193) | 177 (177) | 80 (80)
Solicited Injection Site Swelling (General disorders) | 51 (51) | 69 (69) | 58 (58) | 35 (35)
Irritability (Psychiatric disorders) | 145 (145) | 166 (166) | 166 (166) | 75 (75)
Pyrexia (General disorders) | 25 (25) | 35 (35) | 28 (28) | 22 (22)
Nasopharyngitis (Infections and infestations) | 13 (14) | 19 (19) | 14 (14) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 95 (95) | 101 (101) | 87 (87) | 42 (42)
Somnolence (Nervous system disorders) | 55 (55) | 66 (66) | 54 (54) | 33 (33)
Crying (Psychiatric disorders) | 91 (91) | 91 (91) | 87 (87) | 42 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.